CLINICAL TRIAL: NCT01250223
Title: F2-PROTOCOL: Prospective Collection of Data of Possible Prognostic Relevance in Patients With Follicular Lymphoma
Brief Title: Study of Prognosis of Follicular Lymphoma Through a Prospective Collection of Data (F2-study)
Status: Completed | Type: Observational
Sponsor: Associazione Angela Serra per la ricerca sul cancro (Other)
Collaborators: Fondazione Italiana Linfomi - ETS (Other); The International Non-Hodgkin Lymphoma Prognostic Factor Project (Other)
Responsible Party: Sponsor
Other Study IDs: F2-study
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma, Follicular
Keywords: Lymphoma, Follicular; Prognosis; Progression-Free Survival; Outcome; International Cooperation; Data Collection; Prospective studies; Rare Diseases
MeSH Terms: conditions — Lymphoma, Follicular; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed tissue for central diagnostic pathology review
Oversight: Data Monitoring Committee: No

SUMMARY:
The F2-study is a complement of the previous studies of the Follicular Lymphoma Prognostic Factors Project which permitted the development of the Follicular Lymphoma International Prognostic Index (FLIPI).

The F2-study is designed as a prospective collection of information potentially useful to predict the prognosis of newly diagnosed Follicular Lymphoma patients, and its purposes are to validate the FLIPI and to verify whether a prognostic collection of data would allow the development of a more accurate prognostic index.

DETAILED DESCRIPTION:
So far, in patients with lymphoma a variety of studies aimed at the evaluation of prognosis have been conducted. In particular, different demographic, clinical and biological factors have shown a prognostic role in univariate and multivariate analysis, including age, gender, stage, tumor burden, bone marrow involvement, systemic symptoms, Performance status, serum lactate dehydrogenase (LDH) level, anemia, erythrocyte sedimentation rate (ESR) and beta-2 microglobulin.

The combination of those parameters has allowed the identification of several prognostic scores.

Attempts to define prognosis in follicular lymphomas begun in the late '70s. Then, when in 1993 the International Prognostic Index (IPI) was defined for aggressive lymphomas it was also applied to low-grade lymphomas leading to conflicting results, and the need for a prognostic index specifically designed for follicular lymphomas emerged.

A large study on prognosis in patients with follicular lymphoma was performed by the Italian Lymphoma Intergroup that leaded to the definition of the Italian Lymphoma Intergroup (ILI) score, based on 987 patients (Federico M et al. Blood 2000; 95(3):783-789). In 2004 the Follicular Lymphoma International Prognostic Project allowed the definition of a new score on 4167 pts with follicular lymphoma, the Follicular Lymphoma International Prognostic Index (FLIPI) (Solal-Céligny P et al. Blood 2004;104(5):1258-1265). This score is based on the evaluation of age (younger than 60 years vs 60 years or older), Ann Arbor stage (I-II vs III-IV), number of nodal sites (0-4 vs > 5 or more), Hemoglobin (Hb)level (greater than or equal 12g/dL vs lower than 12g/dL), serum Lactate Dehydrogenase (LDH) (normal vs elevated) and identifies three main groups of patients with different survival:low risk (0-1 factors); intermediate risk (2 factors); high risk (3-5 factors).

Notwithstanding the huge number of patients considered in these studies, all mentioned prognostic scores (IPI, ILI and FLIPI) are based on a retrospective analysis of archive data. This approach can introduce biases that can hamper final results. A first problem is the selection of patients that can be influenced by single institution policy and patient's or physician's related factors. Furthermore, some important variables, such as beta2-microglobulin or Erythrocyte Sedimentation Rate (ESR), that have frequently shown a high prognostic significance in univariate analysis, are hardly included in the final indexes because they are available only in a small number of patients thus loosing their value in multivariate analysis. Then, lacking homogeneous and prospectively defined criteria, retrospective evaluation of some study parameter as for example clinical response cannot be easily defined and all derived endpoints such as Failure Free Survival (FFS)or Progression Free Survival (PFS) may be biased.

Finally the results of a retrospective analysis aiming at the evaluation of survival are dependent on the type of administered treatment and with the recent advent of new drugs such as monoclonal antibodies and purine analogs that can be used also in the elderly patients the role of some established prognostic factor may have changed.

These are the reasons why we thought it would be useful to start a new study based on the prospective registration in a short period of time of patients with follicular lymphoma for whom it would be possible collect an exhaustive set of clinical data and biological information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed follicular lymphoma
* Patients with histologically confirmed diagnosis of follicular lymphoma according to WHO classification (any grade)
* Age over 18
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously-untreated patients with de novo diagnosis of Follicular Lymphoma according to World Health Organization (WHO) classification (grade 1,2,3a,3b)
Sampling Method: Non-Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2003-02; Primary Completion 2008-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5-year

SECONDARY OUTCOMES:
Overall Survival (OS) | 5-year
Event Free Survival (EFS) | 5-year
Treatment Free Survival | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Chair — Dip. Oncologia, Ematologia e Patologie dell'Apparato Respiratorio - Università di Modena e Reggio Emilia, Modena, Italy; Philippe Solal-Céligny, MD, Study Chair — Centre Jean Bernard, Le Mans, France; Armando Lopez-Guillermo, MD, Study Chair — Institut d'Hematologia i Oncologia, Hospital Clinic, Barcelona, Spain; Peter McLaughlin, MD, Study Chair — UT MD Anderson Cancer Ctr, Houston, TX, USA; Umberto Vitolo, MD, Study Chair — Azienda Universitaria Ospedaliera San Giovanni Battista, Torino, Italy; Stefano A. Pileri, MD, Study Chair — Instituto Seragnoli, Unità Operativa di Emolinfopatologia, Università di Bologna, Bologna, Italy
Locations (51):
- United States (3):
  - Northwestern University Feinberg School of Medicine - Department of Hematology/Oncology, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center, Houston, Texas
- Argentina (2):
  - Academia Nacional de Medicina - Oncohematology Department, Instituto de Investigaciones Hematologicas, Buenos Aires
  - Centro de Internacion e Investigacion Clinica "Angelica Ocampo" - Hematologia, Buenos Aires
- Charles University General Hospital - Ist Dept Medicine, Prague, Czechia
- France (6):
  - Centre Hospitalier Universitaire - Hématologie, Besançon
  - Institut Bergonié Comprehensive Cancer Center, Bordeaux
  - Centre Jean Bernard, Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Univeristaire - Hématologie clinique, Nantes
  - Hopital caremeau - Service de Medecine Interne B, Nîmes
  - CHRU Bretonneau - Oncologie medicale, Tours
- Italy (32):
  - Presidio Spedali Civili, Brescia, BS
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Azienda O.U. Vittorio Emanuele-Ferrarotto-S. Bambino, Catania, CT
  - Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, CZ
  - Ospedale Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, FG
  - Ospedale unico Versilia USL 12 - Divisione di Medicina II, DH Oncoematologico, Lido di Camaiore, Lucca
  - Ospedale San Vincenzo - Ematologia e Immunologia, Taormina, Messina
  - Azienda Ospedaliera Ospedali Riuniti Papardo-Piemonte, Messina, ME
  - Istituto Clinico Humanitas, Milan, MI
  - Istituto Scientifico Universitario San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedale Madonna delle Grazie, Matera, Mount
  - Dipartimento di Oncologia, Ematologia e Patologie dell'Apparato Respiratorio, Univ. di Modena e Reggio Emilia - Ematologia, Modena, MO
  - Dipartimento di Oncologia, Ematologia e Patologie dell'Apparato Respiratorio, Univ. di Modena e Reggio Emilia - Medicina Interna, Modena, MO
  - Dipartimento di Oncologia, Ematologia e Patologie dell'Apparato Respiratorio, Univ. di Modena e Reggio Emilia - Oncologia II, Modena, MO
  - Casa di Cura La Maddalena, Palermo, Pa
  - Ospedale civile Guglielmo da Saliceto - Medicina Oncologica ed Ematologica, Piacenza, PC
  - Ospedale Santo Spirito, USL di Pescara - Dipartimento di Oncologia, Pescara, PE
  - Policlinico Monteluce - Divisione di Clinica Medica, Perugia, PG
  - Azienda Ospedaliera Universitaria Pisana - UO di Ematologia, Pisa, PI
  - Fondazione IRCCS Policlinico San Matteo - Clinica Ematologica, Pavia, PV
  - Azienda Ospedaliera S. Carlo - Oncologia Medica, Potenza, PZ
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria, RC
  - Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - Ospedale E. Morelli - Divisione di Medicina Generale, Ematologia, Sondalo, Sondrio
  - Azienda Ospedaliera Universitaria San Giovanni Battista, Torino, TO
  - Policlinico Universitario a gestione diretta - Divisione di Ematologia, Udine, UD
  - Ospedale Civile SS. Giovanni e Paolo - UO di Ematologia, Venezia, VE
  - Azienda Ospedaliera Maggiore della Carità, Novara
  - Azienda Ospedaliera Sant'Andrea - UOC Ematologia, Roma
  - Ospedale Sant'Eugenio - Ematologia, Roma
  - Università la Sapienza, Dip. di Biotecnologie Cellulari ed Ematologia, Sez. Ematologia, Roma
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol - Institut Català d'Oncologia, Badalona
  - Hospital Clinic - Institut d'Hematologia i Oncologia, Barcelona
  - Hospital Universitario Vall de Hebron - Servei d'Hematologia Clinica, Barcelona
  - Institu Catala d'Oncologia - Servei d'Hematologia, Girona
  - Hospital Clinico Universitario, Valencia
- Ospedale S. Giovanni, Bellinzona, Canton Ticino, Switzerland
- Barths and The London NHS Trust, London, United Kingdom

REFERENCES:
- [Result] Federico M, Bellei M, Pro B, Lopez-Guillermo A, Marcheselli L, Trneny M, Soubeyran P, MCLaughlin P, Pileri S, Solal-Céligny P on behalf of the F2 study. Revalidation of FLIPI in patients with Follicular Lymphoma (FL) registered in the F2 study and treated upfront with immunochemotherapy. J Clin Oncol 25(18s), 2007. Abstr 8008.
- [Result] Federico M, Bellei M, Marcheselli L, Luminari S, Lopez-Guillermo A, Vitolo U, Pro B, Martelli M, Soubeyran P, Cortelazzo S, Martinelli G, Pileri S, McLaughlin P, Solal-Céligny P on behalf of International Follicular Lymphoma Prognostic factor Project (IFLPFP) F2-study group. F2 prognostic index. Ann Oncol 19(suppl 4):101-102, 2008. Abstr 058.
- [Result] Federico M, Bellei M, Marcheselli L, Luminari S, Lopez-Guillermo A, Vitolo U, Pro B, Pileri S, Pulsoni A, Soubeyran P, Cortelazzo S, Martinelli G, Martelli M, Rigacci L, Arcaini L, Di Raimondo F, Merli F, Sabattini E, McLaughlin P, Solal-Celigny P. Follicular lymphoma international prognostic index 2: a new prognostic index for follicular lymphoma developed by the international follicular lymphoma prognostic factor project. J Clin Oncol. 2009 Sep 20;27(27):4555-62. doi: 10.1200/JCO.2008.21.3991. Epub 2009 Aug 3. PMID 19652063
- [Result] Solal-Celigny P, Bellei M, Marcheselli L, Pesce EA, Pileri S, McLaughlin P, Luminari S, Pro B, Montoto S, Ferreri AJ, Deconinck E, Milpied N, Gordon LI, Federico M. Watchful waiting in low-tumor burden follicular lymphoma in the rituximab era: results of an F2-study database. J Clin Oncol. 2012 Nov 1;30(31):3848-53. doi: 10.1200/JCO.2010.33.4474. Epub 2012 Sep 24. PMID 23008294